CLINICAL TRIAL: NCT01999985
Title: Phase I Trial Evaluating Safety and Tolerability of the Irreversible Epidermal Growth Factor Receptor Inhibitor Afatinib (BIBW 2992) in Combination With the SRC Kinase Inhibitor Dasatinib for Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase I Trial of Afatinib (BIBW 2992) and Dasatinib in Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17176; BI 1200.166 (Other: Boehringer Ingelheim); BMS CA180-379 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer (NSCLC)
Keywords: Epidermal Growth Factor Receptor (EGFR); Tyrosine kinase inhibitors; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Pleural Diseases; Pleural Neoplasms; Lung Neoplasms; Pleural Effusion; Pleural Effusion, Malignant; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; EGFR mutation; Afatinib; Dasatinib; Carcinoma, Bronchogenic; Gene Mutation; T790M mutation.; Non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Pleural Diseases; Pleural Neoplasms; Pleural Effusion; Pleural Effusion, Malignant; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Carcinoma, Bronchogenic | interventions — Dasatinib; Tyrosine Kinase Inhibitors; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation and Dose Expansion (Experimental): Dose escalation followed by dose expansion. Escalation cohort: Afatinib and Dasatinib. This study is divided into two parts. The first 8 - 18 people will be entered in the first part, called Phase 1A. Then this part will end.
  Expansion cohort:: Afatinib and Dasatinib. The next 20 people will enter into the second part, called Phase 1B.
  Interventions: Drug: Dasatinib - 1A; Drug: Afatinib - 1A; Drug: Dasatinib - 1B; Drug: Afatinib - 1B

INTERVENTIONS:
Drug: Dasatinib - 1A — 1A: Begins Day 8. Level 1 - 100 mg, Level 2 - 100 mg, Level 3 - 140 mg.
  Other Names: SPRYCEL®; BMS-354825; tyrosine kinase inhibitor; SRC Kinase Inhibitor
Drug: Afatinib - 1A — 1A: Begins Day 1. Level 1 - 30 mg, Level 2 - 40 mg, Level 3 - 40 mg.
  Other Names: BIBW 2992; EGFR Inhibitor
Drug: Dasatinib - 1B — In Phase 1B, a mutationally selected 20 participants (total) will be treated at the recommended dose to confirm tolerability and evaluate for early response signal.
Drug: Afatinib - 1B — In Phase 1B, a mutationally selected 20 participants (total) will be treated at the recommended dose to confirm tolerability and evaluate for early response signal.

SUMMARY:
The purpose of this study is to:

* Find out if the study drugs Afatinib and Dasatinib can be safely given together to patients with lung cancer
* Learn how these two drugs work in cancer cells when they are combined
* Learn more about the side effects of these two drugs when combined
* Find the highest doses of the study drugs Afatinib and Dasatinib that can be given safely without causing serious side effects

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically documented Stage IIIB/IV non-small cell lung cancer, or unresectable recurrent disease following locoregional treatment.
* For Phase 1B Extension Only:

  * Either or both of the following: A tumor which harbors an activating Epidermal Growth Factor Receptor (EGFR) - mutation; History of objective response, or stable disease for at least 6 months, after treatment with erlotinib, afatinib, or gefitinib.
  * Either or both of the following: Progression or recurrence of disease after receiving prior continuous gefitinib, afatinib, or erlotinib; A tumor known to harbor a de novo T790M mutation, which is known to confer EGFR TKI resistance.
  * Participants are allowed to have received systemic chemotherapy or investigational therapy in the intervening period prior to trial enrollment
* Capable of giving written informed consent.
* Evaluable disease, as follows: For Phase 1A Dose Escalation: Have the presence of any evaluable disease, including bone metastases, effusion, or cystic metastases. For Phase 1B Extension Only: Have progressive and measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST v 1.1).
* Reproductive potential must be either terminated (by surgery, radiation, or menopause) or attenuated by the use of an approved contraceptive method during and for 3 to 6 months following the study.
* Participant agrees that IV bisphosphonates will be withheld during the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
* Have recovered from prior drug-related toxicity to Grade ≤ 1 Common Terminology Criteria for Adverse Events (CTCAE) v4, within 21 days of initiation of on-study treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at initial enrollment, as assessed by clinician or investigator.

Exclusion Criteria:

* Have previously completed or withdrawn from this study or any other study investigating dasatinib. Prior treatment with other tyrosine kinases, including afatinib, is acceptable.
* Prior recent systemic or investigational therapy within 21 days of initiation of study treatment. An exception is that epidermal growth factor receptor (EGFR) inhibitor may be continued up until 3 days of initiation of study treatment.
* Women who are pregnant or breastfeeding. Women of childbearing potential must have a negative pregnancy test (β-HCG test in urine or serum) prior to commencing study treatment.
* Patients with documented central nervous system or leptomeningeal metastasis (brain metastasis) at the time of study entry. Patients with prior brain metastasis may be considered if they have completed their treatment for brain metastasis and no longer require corticosteroids.
* Patients with disease progression in the central nervous system (CNS) only.
* Serious concomitant disorder, including active bacterial, fungal, or viral infection, incompatible with the study (at the discretion of the principal investigator).
* Uncorrected severe electrolyte disorder, including severe potassium (<3.0 mEq/L) or magnesium ( < 1.0 mEq/L) deficiency.
* Any gastrointestinal disorder with diarrhea as a major symptom, such as Crohn's, or pre-existing chronic diarrhea Common Toxicity Criteria (CTC) Grade ≥ 2 of any etiology. Included are malabsorption disorders that in the opinion of the study physician may affect absorption of either afatinib or dasatinib.
* Prior major surgery or radiation therapy within 14 days of initiation of treatment.
* Electrocardiogram (ECG) abnormalities indicative of arrhythmia (at the discretion of the investigator).
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to enrollment.
* Baseline (< 1 month before treatment) cardiac left ventricular function with resting ejection fraction of less than 50% measured by multigated blood pool imaging of the heart (MUGA scan) or echocardiogram.
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, congenital long QT syndrome, or Torsades de pointes).
* Prolonged QTc interval on pre-entry electrocardiogram (> 470 msec for men and >480 msec for women per American College of Cardiology/American Heart Association [AHA/ACC] 2011 scientific statement).
* History of significant bleeding disorder unrelated to cancer, including diagnosed congenital bleeding disorders (e.g., von Willebrand's disease).
* Patients currently taking drugs that are generally accepted to have a high risk of causing Torsades de Pointes.
* Patients with pre-existing interstitial lung disease (ILD), or pericardial / pleural effusion of grade 2 or higher. Trace pericardial or pleural effusion is acceptable.
* Patients who require chronic oxygen therapy for chronic obstructive pulmonary disease or pleural effusions (malignant or benign).
* Patients requiring comedication with potent P-gp inhibitors (including cyclosporin, azithromycin, erythromycin, ketoconazole, itraconazole, quinidine, phenobarbital salt with quinidine, ritonavir, valspodar, verapamil) or inducers (including rifampicin).
* Known active hepatitis B infection, known active hepatitis C infection, or known HIV carrier.
* Known or suspected active drug or alcohol abuse.
* Known hypersensitivity to afatinib, dasatinib, or the excipients of any of the trial drugs.
* Laboratory exclusion criteria: Absolute neutrophil count (ANC) < 1000 / mm^3, Platelet count < 100,000 / mm^3, Serum creatinine ≥1.5 times the upper normal limit or calculated/measured creatinine Clearance ≤60 mL/min., Total bilirubin ≥1.5 mg/dL (>26 mol/L, SI unit equivalent), Aspartate amino transferase (AST) or Alanine amino transferase (ALT) ≥ 2.5 times the upper limit of normal (if related to liver metastases ≥ five times the upper limit of normal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Creelan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 participants were enrolled at Moffitt Cancer Center from December 2013 to March 2016.
Groups:
- Part 1A Level 1: Participants given 30 mg Afatinib and 100 mg Dasatinib
- Part 1A Level 2: Participants given 40 mg Afatinib and 100 mg Dasatinib
- Part 1B: Participants given Afatinib 30 mg and 100 mg Dasatinib
Period: Overall Study
Arm/Group | Part 1A Level 1 | Part 1A Level 2 | Part 1B
Started | 8 | 3 | 14
Completed | 8 | 3 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- All Participants: All Participants Who Received Study Treatment
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Afatinib (BIBW 2992) in Combination With Dasatinib
Description: The MTD for this combined treatment will be defined as either:
  1. The highest dosage cohort in which six patients had been treated and there were less than two dose limiting toxicities (DLTs) or,
  2. Afatinib at the highest tolerated dose investigated (40 mg by mouth [PO] daily) plus dasatinib at the highest tolerated dose investigated (cohort 3, 140 mg PO daily).
Time Frame: Up to 6 Months
Population: All participants who received at least one dose of Afatinib and Dasatinib.
Measure: Number; unit: mg
Groups:
- Dose Escalation and Expansion: All Participants who received treatment.
Arm/Group | Dose Escalation and Expansion
Number analyzed (Participants) | 25
mg
  Afatinib | 30
  Dasatinib daily | 100

2. Secondary Outcome: Number of Participants With Objective Response
Description: Estimates objective response rate (complete response [CR] and partial response [PR]) in participants with acquired EGFR resistance
Time Frame: Up to 6 Months
Population: All Participants who received treatment.
Measure: Number; unit: participants
Arm/Group | Dose Escalation and Expansion
Number analyzed (Participants) | 25
participants | 0

3. Secondary Outcome: Median Progression Free Survival
Description: Estimate the 6-month progression free survival (PFS) rate in participants with acquired EGFR resistance. Response Criteria for Phase 1B will follow RECIST v.1.1: Progressive Disease (PD) is defined as at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 6 Months
Population: All Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation and Expansion
Number analyzed (Participants) | 25
months | 5.5 [2.6 to 8.5]

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Groups:
- Part 1A Level 1: Participants were given 30 mg Afatinib and 100 mg Dasatinib
- Part 1A Level 2: Participants were given 40 mg Afatinib and 100 mg Dasatinib
Arm/Group | Part 1A Level 1 | Part 1A Level 2 | Part 1B
All-Cause Mortality (participants affected / at risk) | 4/8 | 1/3 | 3/14
Serious Adverse Events (participants affected / at risk) | 5/8 | 2/3 | 9/14
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Level 1 (N=8) | Part 1A Level 2 (N=3) | Part 1B (N=14)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) — Disease progression
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Bronchial hemorrhage
Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Level 1 (N=8) | Part 1A Level 2 (N=3) | Part 1B (N=14)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 3 (7) | 5 (11)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (3) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (2) | 1 (4) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 3 (4)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 2 (2) | 3 (3)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0) | 2 (3)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Weight loss (Investigations) | 1 (1) | 1 (1) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 6 (7)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT01999985/Prot_SAP_000.pdf